CLINICAL TRIAL: NCT01821716
Title: Biological Standardization of Dermatophagoides Pteronyssinus Allergen Extract to Determine the Biological Activity in HEP Units.
Brief Title: Biological Standardization of Dermatophagoides Pteronyssinus Allergen Extract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-PR-PRI-196
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Allergy Dermatophagoides Pteronyssinus; Allergic Rhinitis; Allergic Asthma
Keywords: standardization; skin prick test; inmunotherapy
MeSH Terms: conditions — Dust Mite Allergy; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Three concentrations of Dermatophagoides pteronyssinus allergen extract (10, 1, 0.1 mg/ml)
  Positive control (10 mg/ml histamine dihydrochloride)
  Negative control (glycerinated phenol saline solution)
  Interventions: Biological: Prick test Dermatophagoides pteronyssinus allergen extract

INTERVENTIONS:
Biological: Prick test Dermatophagoides pteronyssinus allergen extract — This is an open, unblinded and non randomized biological as proposed by the Nordic Guidelines.
  Three concentrations of Dermatophagoides pteronyssinus allergen extract, together with a positive and negative control, using 10 mg/ml histamine dichloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. This test will be referred to as the Titrated Skin Prick test.

SUMMARY:
The objective of this study is to determine the biologic activity of a Dermatophagoides pteronyssinus allergen extract in histamine equivalent prick (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

Three concentrations of Dermatophagoides pteronyssinus allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent, appropriately signed and dated by the subject (or legal representative, if applicable).
* Subject can be male or female of any race and ethnic group.
* Age > and =18 years and < and =60 years at the study inclusion day.
* Medical history of allergy with respiratory symptoms (rhinitis and /or rhinoconjunctivitis and/or asthma) to Dermatophagoides pteronyssinus.
* Positive skin prick test with a standardized commercially available preparation of Dermatophagoides pteronyssinus allergen extract. The skin prick test will be considered positive if the test results in a wheal major diameter of at least 3 mm or an area at least 7 mm2. Positive skin prick test results are valid if performed within one year prior to the inclusion of the subject in the study
* A positive test for specific IgE to Dermatophagoides pteronyssinus (CAP-RAST major or equal to 2). IgE results are valid if performed within one year prior to the inclusion of the subject in the study.

Exclusion Criteria:

* Immunotherapy in the past 5 years with a Dermatophagoides pteronyssinus allergen extract or other mites allergen extracts known to interfere with the allergen to be tested, due to a high degree of cross-reactivity.
* Use of drugs that may interfere with the skin reactions (e.g., antihistamines). See Appendix 1 of the protocol.
* Treatment with any of the following medications: oral tricyclic or tetracyclic antidepressants or IMAOs, beta-blockers, chronic use of corticosteroids or use of oral or parenteral corticosteroids in repeated and intermittent patterns (10 mg/daily of prednisone or equivalent).
* Women who are pregnant or period of breastfeeding and women with a pregnancy test positive during the visit 2, prior to the prick test.
* Dermographism affecting the skin area at the test site at either study visit.
* Atopic dermatitis affecting the skin area at the test site at either study visit.
* Urticaria affecting the skin area at the test site at either study visit.
* Diseases of the immune system relevant clinically, both autoimmune and immunodeficiencies.
* Serious diseases not controlled that may increase the risk for the safety of the subjects involved in this study, including, but not limited to the following: heart failure, uncontrolled or severe respiratory diseases,endocrine diseases, clinically relevant kidney or liver diseases or hematological diseases.
* Participation in any other clinical trial within 30 days (or 5 times the biological half-life of the research of the study product, whichever is longer) prior to the inclusion of the subject in this clinical trial.
* Patients with diseases or conditions that limit the use of adrenaline (heart disease, severe hypertension...)
* Severe psychiatric, psychological or neurological disorders
* Abuse of alcohol, drugs or medicines in the previous year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | Test sites should be inspected and recorded 15-20 min after application

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de Denia (Marina Salud), Denia, Alicante
  - Complexo Hospitalario Universitario A Coruña (Hospital Abente y Lago), A Coruña